CLINICAL TRIAL: NCT01687335
Title: Conformity With European Recommendations Concerning the Nutritional Care of the Cancerous Patients Benefiting From a Treatment by Chemotherapy Impact on the Nutritional State and the Quality of Life
Brief Title: Impact on the Nutritional State and the Quality of Life
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00631-40; 2011-11 (Other: AP HM)
Record Dates: First submitted 2011-10-06; First posted 2012-09-18 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cancerous patients: the patients benefiting from treatment by chemotherapy.
  Interventions: Other: answering questionnare in differents time of the treatment

INTERVENTIONS:
Other: answering questionnare in differents time of the treatment

SUMMARY:
The prevalence of malnutrition in cancerous patients varies between 50% and 80%. It is variable in function: the location and the extension of the tumor, of the general state , of age, of the socio-economic class and the pain. The health consequences of a malnutrition are very important: aggravation of the state of health, complications of treatment, hospitalization, alteration of the quality of life and decrease the survival, and the treatment response.

Nutrition being very important in patients, there are recommendations for the nutritional care of these patients, formulated by the European Society for Clinical Nutrition and Metabolism. The investigators do not know to what extent these recommendations are respected in practice and their influence on the nutritional status and the quality of life of patients.

The investigators therefore propose to assess the conformity of the nutritional care patients in clinical practice in relation to the European recommendations and in a second time to assess the influence of this compliance or non-compliance on the nutritional status clinical and biological of cancerous patients under chemotherapy, on their quality of life, on their response to treatment and on their survival.

The investigators will try to identify factors that may be linked to the non-compliance such as the characteristics of the cancer disease, socio-demographic characteristics of the subject and the factors related to the structure in which it is supported.

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old subject in 85 years in the inclusion
* Subject presenting a cancerous pathology requiring a systematic treatment by exclusive chemotherapy for a minimal duration of three months with a plan of 3 cures of chemotherapy with an interval between the cures of 21 days
* Presenting subject one of these 4 cancerous pathologies: cancer of the aéro-digestive ways superiors, sarcomas, colorectal cancers, broncho-lung cancers
* Subject having the capacity of lira and to understand(include) French
* Subject having signed lit(enlightened) consent
* Subject taken care for its cancerous pathology in one of the partner services of the project
* Subject affiliated to the national insurance scheme

Exclusion Criteria:

* Subject having benefited from a major surgical operation in 4 weeks preceding the inclusion
* Subject having benefited from a radiotherapy in two weeks before the inclusion
* Subject minor(miner), pregnant woman, subject incapable to give its consent, subject under supervision(guardianship) - guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancerous patients benefiting from a treatment by chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
quality of life's improvement | 3 YEARS
improvement of treatment effectiveness, | 3 YEARS
improvement of their survival | 3 YEARS

SECONDARY OUTCOMES:
improvement of the screening of the undernutrition | 3 YEARS
the answer to the treatment | 3 years
the estimation of the survival with regard to the nutritional state of the patient. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Salas S, Mercier S, Moheng B, Olivet S, Garcia ME, Hamon S, Sibertin-Blanc C, Duffaud F, Auquier P, Baumstarck K. Nutritional status and quality of life of cancer patients needing exclusive chemotherapy: a longitudinal study. Health Qual Life Outcomes. 2017 Apr 27;15(1):85. doi: 10.1186/s12955-017-0660-6. PMID 28449674